CLINICAL TRIAL: NCT02919124
Title: During Coronary Artery Bypass Surgery. A Feasibility Study.
Brief Title: Epicardial Echocardiography of Coronary Anastomoses Using the Echoclip Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other); Medistim ASA (Industry)
Responsible Party: Principal Investigator, Jan Jesper Andreasen, Professor, MD, PhD, Professor, consultant, Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0089Y
Record Dates: First submitted 2016-09-25; First posted 2016-09-29 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Coronary Arteriosclerosis
Keywords: Coronary artery bypass grafting; Anastomosis; Ultrasonography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Echoclip device (Experimental): Ultrasonography using the echoclip device
  Interventions: Device: Echoclip

INTERVENTIONS:
Device: Echoclip — An ultrasound transducer positioning device, the Echoclip device (Aalborg Hospital, Aalborg,Denmark), which can stabilize the involved part of the myocardium on the beating heart, keep the gel at place, and position the ultrasound transducer correctly for imaging will be used for visualising the coronary bypass anastomoses during surgery

SUMMARY:
The aim of this study is to evaluate whether use of the echoclip device (an ultrasound transducer positioning device which can stabilize the involved part of the myocardium on the beating heart) facilitates imaging of coronary bypass anastomoses during coronary bypass surgery. A total of 100 low risk patients undergoing elective on-pump coronary bypass surgery will be included in the study in order to evaluate if the surgeons can visualize the coronary anastomoses before closure of the sternum. Ultrasonograpic pictures will be analyzed directly peroperatively and electronically post-operatively in order to evaluate if selected areas of the anastomoses can be visualized. Use of the echoclip devise will be considered a success if at least 80% of the anastomoses can be visualized.

DETAILED DESCRIPTION:
The technical quality of coronary artery bypass anastomoses during coronary artery bypass grafting is often evaluated by measuring flow rate in grafts using transit time flowmetry. Unfortunately, flow rate and flow waveform are poor indicators of the anatomy of anastomoses. A better way to evaluate the anatomy of an anastomosis is 3-dimensional imaging. Three problems must be overcome in performing epicardial echocardiography on the beating heart:

1. The transducer must be kept in a steady position relative to the anastomosis for 5 to 10 cardiac cycles to minimize frame-rate variability.
2. Ultrasound gel must be kept in contact with the transducer and the region studied.
3. The transducer must not cause any deformation of the vessels.

The investigators designed an ultrasound transducer positioning device, the Echoclip device (Aalborg Hospital, Aalborg, Denmark), which can stabilize the involved part of the myocardium on the beating heart, keep the gel at place, and position the ultrasound transducer correctly for imaging. The present study is a feasibility study with the aim to evaluate if the echoclip device facilitates imaging of coronary bypass anastomoses during coronary artery bypass surgery in humans to the same degree as was shown in animal studies. Ultrasonography will be used for visualizing all coronary anastomoses during 100 elective low-risk (logistic II EuroSCORE <6) on-pump coronary artery bypass procedures. It will be registered if the heel, the central portion and the toe of the anastomosis can be visualized in end-to-side and side-to-side anastomoses.Use of the echoclip devise will be considered a success if at least 80% of all parts of the anastomoses can be visualized either directly or by electronic reading using a special developed algorithm that may identify the inner border of the anastomoses.

ELIGIBILITY:
Inclusion Criteria:

* Elective on-pump coronary artery bypass surgery
* Surgery planned to be performed by specialist in cardiac surgery.
* Logistic euroSCORE II <6%.
* Must be able to read and understand the Danish
* Written informed acceptance to participate

Exclusion Criteria:

* Planned off-pump surgery.
* Peroperativ conversion to off-pump surgery.
* Logistic EuroSCORE II ≥ 6.
* The patient do not understand written or spoken Danish.
* Surgery within 24 hours after admittance to hospital
* Patients in whom the surgeon wants to end the surgery in a hurry due to e.g. hemodynamic problems or peroperative complications.
* The surgeon is not a specialist in cardiac surgery, e.g. surgeon in training.
* Pregnant or brest feeding patient.
* No written acceptance to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-09; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of periferal coronary artery bypass anastomotic structures | Peroperative
  Ultrasonographic images of periferal coronary artery bypass anastomoses will be studied in order to evaluate if the area of anastomotic structures from various locations of the anastomoses (heel, central portion and the to toe) can be visualized directly on the screen using the echoclip device.

SECONDARY OUTCOMES:
Automatic quality control of periferal coronary artery bypass anastomotic structures | Peroperative
  To quantify the anastomotic quality from epicardial utrasound images obtained peroperative, the area of anastomotic structures from various locations of the anastomoses (heel, central portion and the to toe) will be meassured using an automatic anastomosis segmentation algorithm to extract the area of the anastomotic structures. The ultrasound images obtained peroperative will be analyzed in the Laboratory when 50 patients and 100 patients have been included in the study, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jan J Andreasen, MD, PhD, Principal Investigator — Aalborg University Hospital and Aalborg University
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are available for Monitor

REFERENCES:
- [Result] Staalsen NH, Kjaergaard B, Andreasen JJ. A new technique facilitating intraoperative, high-frequency echocardiography of coronary bypass graft anastomoses. J Thorac Cardiovasc Surg. 2011 Jan;141(1):295-6. doi: 10.1016/j.jtcvs.2009.11.074. No abstract available. PMID 21168035
- [Derived] Jorgensen AS, Andersen MS, Ostergaard LR, Schmidt SE, Nohr D, Andreasen JJ. A laboratory feasibility study using a computer algorithm for anastomosis segmentation of epicardial ultrasonography images from distal coronary artery bypass anastomoses. J Cardiothorac Surg. 2025 Jan 6;20(1):34. doi: 10.1186/s13019-024-03187-8. PMID 39762954
- [Derived] Andreasen JJ, Nohr D, Jorgensen AS, Haahr PE. Peroperative epicardial ultrasonography of distal coronary artery bypass graft anastomoses using a stabilizing device. A feasibility study. J Cardiothorac Surg. 2020 Jan 8;15(1):3. doi: 10.1186/s13019-020-1057-x. PMID 31915030
- [Derived] Andreasen JJ, Nohr D, Jorgensen AS. A case report on epicardial ultrasonography of coronary anastomoses using a stabilizing device without the use of ultrasound gel. J Cardiothorac Surg. 2019 Mar 13;14(1):59. doi: 10.1186/s13019-019-0882-2. PMID 30866994